CLINICAL TRIAL: NCT02510144
Title: Adjusting Skin Prep to Decrease Risk of P. Acnes Related Shoulder Infection
Brief Title: Skin Prep to Reduce Postoperative Shoulder Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mohit N. Gilotra, Assistant Professor of Orthopaedics, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00064296
Record Dates: First submitted 2015-07-23; First posted 2015-07-29 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Shoulder Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine (Active Comparator): A preoperative Chlorhexidine gluconate solution 4.0% (i.e Hibiclens)
  Interventions: Drug: Skin Prep Chlorhexidine
- Benzoyl Peroxide (Experimental): A preoperative 5% benzoyl peroxide wash prep (i.e. Brevoxyl-4 and Brevoxyl-8)
  Interventions: Drug: Skin Prep Benzoyl Peroxide

INTERVENTIONS:
Drug: Skin Prep Chlorhexidine — 3 day preoperative skin prep prior to surgery
  Arms: Chlorhexidine
Drug: Skin Prep Benzoyl Peroxide — 3 day preoperative skin prep prior to surgery
  Arms: Benzoyl Peroxide

SUMMARY:
Propionibacterium acnes is the most common pathogen identified from a surgical site infection in the shoulder. Standard skin preps do not prevent this type of infection. Patients will undergo either a chlorhexidine or benzoyl peroxide prep in days leading up to surgery. Bacterial burden will be determined at the time of surgery.

DETAILED DESCRIPTION:
After surgical posting, patients will be randomized to chlorhexidine or benzoyl peroxide group. The solutions used will be 5% benzoyl peroxide emollient foam and 4% chlorhexidine gluconate skin cleanser. Participants will be instructed to conduct skin wash using the appropriate solution in the shower over the operative shoulder and axilla for three mornings prior to surgery (pre op day -2, pre op day -1, and morning of surgery). Specific instructions will include leaving the solution on the skin for three minutes and avoiding contact with eyes, ears, and mouth. Proper technique will be demonstrated at time of patient recruitment and given as a handout with the wash solution provided. A reminder phone call will occur two days before surgery to remind patients of proper procedure to improve compliance. On the day of surgery, patients be interviewed about pre-operative compliance.

On the day of surgery, two cultures will be taken in three separate sites on both shoulders (anterior, lateral, and posterior) using a detergent scrub technique, the current dermatologic standard for biopsy of the deep sebaceous glands. (3,11) This procedure is typically performed on the skin of awake patients and causes minimal pain and skin irritation. Cultures will be evaluated in our lab. We will also test for hemolysis as a possible indicator of a more virulent strain in the literature.

The research team may take photos of the shoulder skin being swabbed. Photos will not include the facial or defining characteristics. Photos may be taken either in the clinic at time of recruitment or in the operating room when samples are being taken.

Inclusion criteria: all patients undergoing open shoulder surgery or shoulder arthroscopy. Exclusion criteria: anyone with a history of allergic reaction to chlorhexidine or benzoyl peroxide. Anyone with a history of previous shoulder infection, current open skin lesions around the shoulder or the use of current anti-acne medications around the shoulder.

Healthy volunteer portion: Healthy volunteers will respond to the study from fliers on campus. A cotton swab test on both shoulders will be performed prior to any treatment. If a threshold of P. Acnes is met (>1000 Colony Forming Units (CFUs)) then volunteers will be randomized to the same two groups and retested after three days of unilateral treatment. Finally, volunteers will undergo repeat cotton swab testing one week after 3 day wash was finalized.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Indicated for shoulder surgery

Exclusion Criteria:

* History of previous shoulder infection
* Allergy to Chlorhexidine or benzoyl peroxide
* Current use of anti-acne medicine around the shoulder
* Patient is pregnant or concerned about pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Midtown Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chlorhexidine | Benzoyl Peroxide
Started | 39 | 41
Completed | 39 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine | Benzoyl Peroxide | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Full Range); unit: years] | 51 [18 to 88] | 51 [23 to 77] | 51 [18 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 19 | 18 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80
BMI [Mean (Full Range); unit: kg/m^2] | 30.2 [20.0 to 47.4] | 30.7 [18.0 to 45.8] | 30.5 [18.0 to 47.4]
Active smokers [Count of Participants; unit: Participants] | 10 | 13 | 23
Diabetes [Count of Participants; unit: Participants] | 8 | 8 | 16
Arthroplasty cases [Count of Participants; unit: Participants] | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Skin Swab and Culture With Colony Forming Units (CFUs)
Description: Preoperative Cutibacterium acnes shoulder burden. Skin cultures of both shoulders were obtained via a detergent scrub technique the day of surgery at anterior, lateral, and posterior sites and the axilla.
Time Frame: At time of surgery
Population: 8 samples/skin cultures were obtained from each participant; 4 from each shoulder. The contralateral shoulder was the control.
Measure: Number; unit: negative skin cultures
Units Other Than Participants: skin cultures
Arm/Group | Chlorhexidine | Benzoyl Peroxide
Number analyzed (Participants) | 39 | 41
Number analyzed (skin cultures) | 156 | 164
negative skin cultures
  Intervention | 39 | 51
  Control | 35 | 22
Statistical Analysis 1: Comparison: Chlorhexidine; Negative cultures were compared on the treated side vs the non-treated side; Test type: Superiority; p = 0.68, t-test, 2 sided
Statistical Analysis 2: Comparison: Benzoyl Peroxide; Negative cultures were compared on the treated side versus the non-treated side; Test type: Superiority; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Surgical Site Infection That Requires Antibiotics
Description: Cultures were evaluated in our lab and also tested for hemolysis as a possible indicator of a more virulent strain in the literature.
Time Frame: At one year
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine | Benzoyl Peroxide
Number analyzed (Participants) | 39 | 41
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Chlorhexidine | Benzoyl Peroxide
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02510144/Prot_SAP_000.pdf